CLINICAL TRIAL: NCT05868837
Title: Single-cell Deep Phenotyping of B Lymphocytes to Personalize Immunotherapy in Patients With Myasthenia Gravis: Clinical Trial to Evaluate the Efficacy and Safety of Rituximab in Generalized AChR-antibody Positive Myasthenia Gravis
Brief Title: Rituximab EfFicacy IN MyasthEnia Gravis (REFINE)
Acronym: REFINE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3916
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2024-09

CONDITIONS: Myasthenia Gravis, Generalized
MeSH Terms: conditions — Myasthenia Gravis | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rituximab (Experimental): Rituximab will be provided in 500mg/50ml vials; excipients include sodium chloride, tri-sodium citrate dihydrate, polysorbate 80, water for injections. Two vials will be diluted in 500 ml of sodium chloride 0,9% to reach a concentration of 2mg/ml. Rituximab will be administered intravenously in two 1000 mg infusions, with two weeks distance between the first and the second infusion.
  Interventions: Drug: Rituximab
- Placebo (Placebo Comparator): Placebo will consist of 500 ml flacons of sodium chloride 0,9%.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rituximab — Rituximab 1000 mg IV on RCP days 1 and 15
  Other Names: MabThera; Rituxan
  Arms: Rituximab
Other: Placebo — Placebo 1000 mg IV on RCP days 1 and 15
  Arms: Placebo

SUMMARY:
The primary objective of this phase III trial is to investigate if Rituximab can reduce patients' functional impairment caused by MG. The secondary objectives of this trial are to assess whether treatment with rituximab in patients with MG will:

* Allow faster and greater corticosteroid tapering
* Reduce the frequency of exacerbations
* Improve quality of life
* Offer an acceptable safety and tolerability profile.

ELIGIBILITY:
Inclusion Criteria:

a. Positive serologic test for anti-AChR or anti-MuSK antibody titers as confirmed at screening (one retest allowed), and

At least one of the following:

i)-History of abnormal neuromuscular transmission test results demonstrated by single- fiber electromyography or repetitive nerve stimulation; or ii)-History of positive anticholinesterase test (eg, edrophonium chloride test); or iii)-Patient demonstrated improvement in MG signs on oral cholinesterase inhibitors, as assessed by the treating physician; or iv)-Clinical syndrome consistent with a diagnosis of MG, and not otherwise explained by another condition. c. MGFA Clinical Classification Class II, III, or IV at the time of screening and randomization.

d. MG-ADL score of 5 or greater at screening and at randomization with > 50% of this score attributed to non-ocular items. e. QMG score of 11 or greater at screening and at randomization. f. Willing and able to comply with the protocol, complete study assessments, and return for follow- up visits.

g. Females of childbearing potential who are sexually active with a non-sterilized male partner must use at least one highly effective contraception method (Table 1) from the time of screening and for 12 months after the final dose of IP. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception. h. Females of childbearing potential are defined as those who are not surgically sterile (ie, bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or those who are not postmenopausal (defined as 12 months with no menses without an alternative medical cause).

i. Non-sterilized males who are sexually active with a female partner of childbearing potential must use a condom from Day 1 for the duration of the study and for 3 months after the last dose of IP. Because male condom is not a highly effective contraception method, it is strongly recommended that female partners of a male study subject also use a highly effective method of contraception throughout this period.

Exclusion Criteria:

1. Any condition that, in the opinion of the Investigator, would place the patient at unacceptable risk of complications, interfere with evaluation of the IP, or confound the interpretation of patient safety or study results.
2. Lactating or pregnant females, or females who intend to become pregnant anytime from signing the informed consent form (ICF) throughout the RCP plus 6 months following last dose of IP.
3. History of drug or alcohol abuse within < 1 year prior to screening, or any condition associated with poor compliance as judged by the Investigator.
4. Site staff and their family members.
5. Currently committed to an institution by way of official or judicial order.
6. Subjects diagnosed with congenital myasthenic syndromes.
7. Known immunodeficiency disorder, including human immunodeficiency virus (HIV) infection.
8. Thymectomy within ≤ 12 months prior to baseline (Day 1) visit or planned thymectomy during the duration of the RCP.

10. Receipt of the following medications or treatments at any time prior to randomization:

1. Alemtuzumab (Lemtrada®, Campath®)
2. Total lymphoid irradiation
3. Bone marrow transplant
4. T-cell vaccination therapy
5. Natalizumab (Tysabri®) 10. Receipt of ANY immunosuppressive treatment (excluding corticosteroids) at ANY time prior to randomization (such as Azathioprine, Mycophenolate mofetil or Mycophenolic acid, Cyclosporine (except eye drop), Tacrolimus (except topical), Methotrexate, Cyclophosphamide, Tocilizumab (Actemra®), Belimumab (Benlysta®), Eculizumab (Soliris®), rituximab (MabThera®, Rituxan®), ocrelizumab (Ocrevus®), ofatumumab (Arzerra®), obinutuzumab (Gazyva®), inebilizumab, or any experimental B-cell depleting agent) 11. Receipt within the 4 weeks prior to Day 1:

a. Intravenous immunoglobulin (IVIg) b. Plasma exchange (PLEX) treatment 12. Current use of:

1. Prednisone < 20 mg/day or < 40 mg over a 2-day period (or equivalent dose of other corticosteroids)
2. Pyridostigmine > 480 mg/day or unstable dose in the 2 weeks prior to Day 1 13. Concurrent/previous enrollment in another clinical study involving an investigational treatment within 4 weeks or 5 half-lives of the investigational treatment, whichever is longer, prior to Day 1.

   14. Receipt of a live attenuated vaccine within 4 weeks prior to randomization. Administration of inactivated (killed) vaccines is acceptable. 15. History of severe allergic or anaphylactic reactions to biologic agents or known allergy to any component of the IP formulation. 16. History of recurrent significant infections (eg, requiring hospitalization or IV antibiotics).

   17. Within 2 weeks prior to the screening visit: clinically significant active infection requiring antimicrobial medication but allowing chronic nail infections. 18. Unresected thymoma (Note: subjects with a benign thymoma resected > 1 year prior to screening may enroll. Benign is defined as no known metastases and no extension into or beyond the capsule on pathological examination. Imaging to evaluate for thymoma must have been performed prior to randomization per standard of care). 19. History of cancer, except for the following:

a. In situ carcinoma of the cervix treated with apparent success with curative therapy for > 12 months prior to screening b. Cutaneous basal cell or squamous cell carcinoma treated with apparent success with curative therapy for > 12 months prior to screening c. Prostate cancer treated with radical prostatectomy or radiation therapy with curative intent > 3 years prior to screening and without known recurrence or current treatment d. Malignant thymoma (i.e. Masaoka stage ≥ IIa) resected > 5 years prior to screening with no evidence of active disease and no therapy received over the previous 5 years. Imaging to evaluate for thymoma must have been performed prior to randomization per standard of care 21. Spontaneous or induced abortion, still or live birth, or pregnancy ≤ 4 weeks prior to screening.

22. Any of the following laboratory abnormalities at screening (one repeat test may be conducted to confirm results prior to randomization within the same screening period):

a. Elevated liver enzymes (aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 × upper limit of normal (ULN)). b. Total bilirubin > 1.5 × ULN (unless due to Gilbert's syndrome) c. Estimated glomerular filtration rate (eGFR) < 45 mL/min/1.73 m2 d. CD19+ B-cell count < 40 cells/μL e. Absolute neutrophil count (ANC) < 1.2 × 103 cells/μl f. Platelet count < 75,000/μL (or < 75 × 109/L) g. Hemoglobin < 8.0 g/dL h. Total immunoglobulin < 600 mg/dL 23. Positive test for chronic hepatitis B infection at screening, defined as either (1) positive hepatitis B surface antigen (HBsAg) or (2) a positive hepatitis B core antibody (anti-HBc) PLUS negative hepatitis B surface antibody (anti-HBs). Note: Subjects with a positive anti-HBs only, or a positive anti-HBc plus positive anti-HBs and negative HBsAg, are eligible to enroll. 24. Positive test for hepatitis C virus antibody. 25. Positive HIV test. 26. Blood transfusion within 4 weeks prior to screening or during the screening period.

27. Inability to read. 28. History of active or latent tuberculosis (TB), or a positive QuantiFERON®-TB Gold test at screening, unless treatment for tuberculosis was completed per local guidelines. Subjects with latent TB or a positive QuantiFERON®-TB Gold test who are actively on anti-TB treatment can enroll if they have completed at least 1 month of anti-TB treatment and intend to complete the full course of anti-TB treatment. Subjects with an indeterminate QuantiFERON®-TB Gold test result can enroll if a repeat QuantiFERON®-TB Gold is negative or a tuberculin skin test is negative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
To assess whether rituximab can reduce MG-related functional impairment. | 12 weeks
  Change from baseline in Quantitative Myasthenia Gravis Score (QMG) at week 12 (3 months) of the RCP.
  QMG score 0 - 39 A higher score means a worse outcome

SECONDARY OUTCOMES:
To evaluate the effect of rituximab on corticosteroid usage. | 48 weeks
  Change in corticosteroid dosage from week 12 to the end of the RCP.
To evaluate the effect of rituximab on MG-related disability. | 12 weeks
  Change from baseline in Myasthenia Gravis Activities of Daily Living (MG-ADL) score at week 12.
  MG-ADL score 0 - 24 A higher score means a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Iorio, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Policlinico A. Gemelli IRCCS, Roma, Italy